CLINICAL TRIAL: NCT04016753
Title: The Effect of BMS-986256 on the Pharmacokinetics of a Combined Oral Contraceptive (Ethinyl Estradiol/Norethindrone) in Healthy Female Participants
Brief Title: A Study Measuring the Effectiveness of BMS-986256 Combined With Oral Contraceptive in Healthy Female Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IM026-021
Record Dates: First submitted 2019-06-26; First posted 2019-07-11 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: Healthy Participants
MeSH Terms: interventions — norethindrone acetate, ethinyl estradiol, ferrous fumarate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Monotherapy (Experimental)
  Interventions: Drug: BMS-986256; Drug: Loestrin

INTERVENTIONS:
Drug: BMS-986256 — 30 mg(6ml)
Drug: Loestrin — 1.5 mg Norethindrone and 30ug ethinyl estradiol

SUMMARY:
A comparative study of BMS-986256 with a combined oral contraceptive in healthy female participants to determine the effectiveness when taken together

ELIGIBILITY:
Inclusion Criteria:

* Participants must be a non- smoking genetically female, who has normal renal function, willing to use Loestrin, and of childbearing Potential with intact ovarian function.
* Participants must be healthy, defined as having no clinically significant active or ongoing medical condition Weighing less than or equal to 50 kg and a body mass index between 18.0 and 32.0kg inclusive at screening.
* Participant must have a negative QuantiFeron- TB Gold test at screening and have a normal pap smear result within 3 years.

Exclusion Criteria:

* Participants who are involuntarily incarcerated, have a significant Chronic medical illness or a history of relevant drug allergy to immunologic or related compounds.
* Any serious bacterial, fungal, or viral infection within 3 months or a history of recurrent or chronic infection or Risk for TB.
* A history of any medical condition specifically related to the use of hormonal contraceptives as well as an average intake of more than 21 units of alcohol per week.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma Concentration (Cmax) of Norethindrone (NET) | Day 21 of cycle 1 and cycle 2 (each cycle is 28 days)
Area under the plasma concentration-time curve over the dosing interval AUC(TAU) of NET | Day 21 of cycle 1 and cycle 2 (each cycle is 28 days)
Maximum observed plasma Concentration (Cmax) of Ethinyl Estradiol (EE) | Day 21 of cycle 1 and cycle 2 (each cycle is 28 days)
Area under the plasma concentration-time curve over the dosing interval AUC(TAU)of (EE) | Day 21 of cycle 1 and cycle 2 (each cycle is 28 days)

SECONDARY OUTCOMES:
Incidence of Adverse Events (AEs) | Up to 28 weeks
Incidence of Serious Adverse Events (SAEs) | Up to 28 weeks
Serology clinical lab assessment of blood | up to 28 weeks
Hematology clinical lab assessments of blood | up to 28 weeks
Urinalysis clinical lab assessment | up to 28 weeks
Vital signs of blood pressure | up to 28 weeks
Vital signs of body temperature | up to 28 weeks
Vital signs of respiratory rate | up to 28 weeks
Number of Participants with abnormal physical examination findings | up to 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Altasciences Los Angeles (Formerly WCCT Global), Cypress, California, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm